CLINICAL TRIAL: NCT06061029
Title: A Brief Yoga- and Mindfulness-Based Psychoeducation Program for Women Who Have Experienced Domestic Violence: A Randomized Control Trial Study
Brief Title: Brief Yoga and Mindfulness for Women Who Have Experienced Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Navidreza Hosseinzadeh ASL, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/06
Record Dates: First submitted 2023-09-19; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Domestic Violence
Keywords: Brief yoga and mindfulness; online psychoeducation; self-compassion; rumination; domestic violence; psychological health
MeSH Terms: conditions — Rumination Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga- and Mindfulness-Based Psychoeducation Program Group (Experimental)
  Interventions: Behavioral: Brief Yoga- and Mindfulness-Based Psychoeducation Program
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Brief Yoga- and Mindfulness-Based Psychoeducation Program — A unique mindfulness psychoeducation program incorporating features of Hatha yoga and mindfulness-based cognitive therapy, plus the main concepts of self-compassion
  Arms: Yoga- and Mindfulness-Based Psychoeducation Program Group

SUMMARY:
This study aimed to examine the effectiveness of a brief yoga- and mindfulness-based psychoeducation program and its working mechanisms in improving psychological health parameters (depression, anxiety, and stress) among women who have experienced domestic violence (DV).

In a randomized controlled trial, 51 DV-victimized women were assigned to an intervention group (n = 27) or a waitlist control group (n = 24). The intervention was a five-week yoga- and mindfulness-based psychoeducation program.

The researchers planned to provide support for the effectiveness of a brief yoga- and mindfulness-based psychoeducation program for improving the psychological health of DV-victimized women. Self-compassion and rumination were hypothesized as working mechanisms underlying the intervention's success.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study required participants to be women aged 18 years or older who had experienced domestic violence in the previous 12 months but were no longer in an ongoing domestic violence situation. Additionally, participants needed to have secure access to a smartphone or a laptop / Personal Computer.

Exclusion Criteria:

* Refusal to give consent or missing more than one session of the psychoeducation program were the exclusion criteria. The individuals who met the absence criterion were still able to continue the rest of the sessions; however, their questionnaires were not included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales-21 | 6 weeks
  To measure the occurrence of symptoms associated with depression, anxiety, and stress. In this scale, higher scores mean higher depression, anxiety, or stress.
The Self-Compassion Scale-Short Form | 6 weeks
  To measure self-compassion level. In this scale higher scores mean better/higher self-compassion.
The Brief State Rumination Inventory | 6 weeks
  To measure rumination level. In this scale higher scores mean higher rumination.

CONTACTS AND LOCATIONS:
Locations (1):
- Navidreza Hosseinzadeh Asl, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data supporting the results of this study can be obtained from the corresponding author upon a reasonable request. The data cannot be made publicly accessible due to their containing sensitive information that could potentially breach the confidentiality of research participants. Nonetheless, the authors are dedicated to providing access to the data for interested researchers in a responsible and transparent manner, while adhering to all applicable ethical and legal standards.